CLINICAL TRIAL: NCT06268366
Title: Effects of Exercise-Based Interventions on Symmio Self-Movement Screen Scores in Untrained Adults_ A Randomized Controlled Trial
Brief Title: Effects of Exercise-Based Interventions on Symmio Self-Movement Screen
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Evansville (Other)
Responsible Party: Principal Investigator, Kyle Matsel, Associate Professor, University of Evansville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UEvansville
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Movement Disorders
Keywords: Symmio Self-Movement Screen; Intervention; Wellness
MeSH Terms: conditions — Movement Disorders | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The primary investigators and statisticians will be blinded to the group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in the control group will not receive any exercise interventions. Participants in the control group will receive their individualized corrective exercises program following completion of the research study following the 10 week follow up.
- Exercise Group (Experimental): Participants in the intervention will be assigned three corrective exercises based on their greatest movement pattern deficit as advised by the Symmio application. Participants in the intervention group will follow the exercise and educational guidance provided by the Symmio application including adjustment of exercises and reviewing educational materials.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Three exercises consisting of stretching and strengthening specific to the movement pattern dysfunction scored by Symmio will be prescribed to the participants. The exercises are standardized and assigned within the Symmio application with video instruction and guidance.
  Arms: Exercise Group

SUMMARY:
Musculoskeletal screening for physical risk factors requires equipment and a trained healthcare or fitness professional to perform and interpret the scoring so that appropriate exercise interventions can be prescribed. However, barriers such as healthcare costs and accessibility, low perceived need to seek medical care, and previous unfavorable evaluation of seeking medical care are associated with healthcare avoidant behaviors. This research aims to explore the effectiveness of the Symmio Self-Screen application to generate specific exercise interventions to address an individual's associated physical risk factors. The ability of the Symmio application to prescribe a targeted exercise program which can reduce asymmetries, improve movement quality, and enhance overall function is unknown. Therefore, the purpose of this study is to determine the effectiveness of the Symmio application in designing individualized exercise interventions which target the unique movement limitations and asymmetries in adults.

DETAILED DESCRIPTION:
Musculoskeletal disorders (MSDs) are currently the largest category of workplace injuries, accounting for 30% of all workers compensation costs, and are on the rise. Globally, MSDs are also on the rise in the general adult population with 1 in 3 adults with some report of an MSD. In the United States, MSDs are even more prevalent with 1 in 2 adults presenting with a musculoskeletal disorder. The financial implications of MSDs are extensive. In the United States, annual healthcare costs associated with MSDs have surpassed $380 billion. Among the most prevalent musculoskeletal disorders were low back pain and neck pain, accounting for a 6.7% spending increase annually from 1996 to 2016.

Increased physical activity is a proven way to decrease the prevalence of MSK risk factors and improve overall health. However, trends suggest MSK disorders and physical inactivity are becoming more prevalent. Generalized exercises programs may not be specific enough to effectively manage physical risk factors. Furthermore, starting a general exercise program to address the adverse effects of inactivity is now considered a risk factor for the development of an MSD. This is likely due to inappropriate functional foundations which cannot withstand the rigors of moderate to high level physical activity. Identification and mitigation of physical risk factors could establish a better movement foundation and provide individuals the durability to achieve their long-term fitness goals.

Several musculoskeletal movement screens exist which can identify physical risk factors and are associated with injury prediction. The Functional Movement Screen (FMS™) and Y-Balance Test - Lower Quarter (YBT-LQ™) are reliable, movement-based tests which can identify modifiable risk factors related to mobility and motor control deficits. However, both the FMS™ and YBT-LQ™ require equipment and are administered by a trained healthcare or fitness professional. Furthermore, the professional is required to interpret the scoring and to prescribe appropriate exercise interventions to improve specific movement limitations or asymmetries. However, barriers such as healthcare costs and accessibility, low perceived need to seek medical care, and previous unfavorable evaluation of seeking medical care are associated with healthcare avoidant behaviors.

The Symmio Self-Screen (Symmio) is a downloadable application developed to be a user-friendly and cost-effective tool for the early identification of physical risk factors that may lead to MSK injuries. The Symmio Self-Screen application provides step by step directions to screen for basic movement pattern limitations and asymmetries. Recently, the Symmio application was found to be highly reliable and valid when used as a self-screening tool to assess MSK risk factors. The simplistic scoring criteria and video guided instructions offered through the application allows for untrained adults to self-score their own movement patterns similarly to a trained healthcare provider. Additionally, the accuracy of Symmio to identify painful movement, movement dysfunction on the FMS™, and dynamic balance deficits on the YBT-LQ™ was 0.74, 0.73, 0.69, respectively. Information gained from this screening approach could allow the general population to self-screen and monitor for the development of physical risk factors and intervene with targeted exercises interventions prior to the onset of symptoms or injury.

To date, the effectiveness of the Symmio Self-Screen application to generate specific exercise interventions to address an individual's associated physical risk factors has not been explored. The ability of the Symmio application to prescribe a targeted exercise program which can reduce asymmetries, improve movement quality, and enhance overall function is unknown. Therefore, the purpose of this study is to determine the effectiveness of the Symmio application in designing individualized exercise interventions which target the unique movement limitations and asymmetries in adults. It is hypothesized that individuals who receive specific exercise interventions recommended by the Symmio application will have less asymmetries, improve performance on the Symmio Self-Movement Screen, and better function compared to a control group which will not receive individualized exercises.

ELIGIBILITY:
Inclusion Criteria:

* Willing participants between the ages of 18 to 65 years of either sex
* At least 1 less than optimal movement pattern scored on the Symmio Self-Movement Screen.

Exclusion Criteria:

* Optimal scores on all Symmio movement patterns
* Current lower extremity injury
* Lower extremity or upper extremity amputation
* Lack of medical clearance from physician/primary care to participate in exercise
* Undergoing current medical treatment for musculoskeletal injury
* Concussion within the past 3 months
* Inability to read and comprehend English.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Symmio Self-Movement Screen | Baseline, 3 weeks, 6 weeks, and 10 weeks
  Each participant will have access to the Symmio application via cell phone or tablet and will complete the self-screen as directed by the video and verbal guidance provided in the application. Participants will self-score themselves on the Symmio movements and record their results into both the application and on the data collection form.

SECONDARY OUTCOMES:
Global Rating of Change | 3 weeks, 6 weeks, and 10 weeks
  Each participant's global rate of change (GROC) will be evaluated at each follow-up time point. GROC ratings that positively change categories toward improvement will be considered positive outcomes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alemany JA, Bushman TT, Grier T, Anderson MK, Canham-Chervak M, North WJ, Jones BH. Functional Movement Screen: Pain versus composite score and injury risk. J Sci Med Sport. 2017 Nov;20 Suppl 4:S40-S44. doi: 10.1016/j.jsams.2017.08.001. Epub 2017 Aug 23. PMID 28919122
- [Background] Bonazza NA, Smuin D, Onks CA, Silvis ML, Dhawan A. Reliability, Validity, and Injury Predictive Value of the Functional Movement Screen: A Systematic Review and Meta-analysis. Am J Sports Med. 2017 Mar;45(3):725-732. doi: 10.1177/0363546516641937. Epub 2016 Jul 21. PMID 27159297
- [Background] Booth FW, Roberts CK, Laye MJ. Lack of exercise is a major cause of chronic diseases. Compr Physiol. 2012 Apr;2(2):1143-211. doi: 10.1002/cphy.c110025. PMID 23798298
- [Background] Booth FW, Roberts CK, Thyfault JP, Ruegsegger GN, Toedebusch RG. Role of Inactivity in Chronic Diseases: Evolutionary Insight and Pathophysiological Mechanisms. Physiol Rev. 2017 Oct 1;97(4):1351-1402. doi: 10.1152/physrev.00019.2016. PMID 28814614
- [Background] Butler RJ, Contreras M, Burton LC, Plisky PJ, Goode A, Kiesel K. Modifiable risk factors predict injuries in firefighters during training academies. Work. 2013 Jan 1;46(1):11-7. doi: 10.3233/WOR-121545. PMID 23324700
- [Background] Dieleman JL, Cao J, Chapin A, Chen C, Li Z, Liu A, Horst C, Kaldjian A, Matyasz T, Scott KW, Bui AL, Campbell M, Duber HC, Dunn AC, Flaxman AD, Fitzmaurice C, Naghavi M, Sadat N, Shieh P, Squires E, Yeung K, Murray CJL. US Health Care Spending by Payer and Health Condition, 1996-2016. JAMA. 2020 Mar 3;323(9):863-884. doi: 10.1001/jama.2020.0734. PMID 32125402
- [Background] Hart, P. D. (2017). Epidemiology of Exercise-Related Injuries Presenting to U.S. Emergency Departments: 10-year Trends. Journal of Physical Fitness, Medicine & Treatment in Sports, 1. https://doi.org/10.19080/JPFMTS.2017.01.555562
- [Background] Kiesel KB, Butler RJ, Plisky PJ. Prediction of injury by limited and asymmetrical fundamental movement patterns in american football players. J Sport Rehabil. 2014 May;23(2):88-94. doi: 10.1123/jsr.2012-0130. Epub 2013 Nov 14. PMID 24225032
- [Background] March L, Smith EU, Hoy DG, Cross MJ, Sanchez-Riera L, Blyth F, Buchbinder R, Vos T, Woolf AD. Burden of disability due to musculoskeletal (MSK) disorders. Best Pract Res Clin Rheumatol. 2014 Jun;28(3):353-66. doi: 10.1016/j.berh.2014.08.002. Epub 2014 Nov 18. PMID 25481420
- [Background] Matsel K, Kirsch J, Netelbeek T, Rodriguez R, Velic E, Schwartzkopf-Phifer K. Self-Movement Screening using the Symmio Application is Reliable and Valid for Identifying Musculoskeletal Risk Factors. Int J Sports Phys Ther. 2023 Apr 1;18(2):439-449. doi: 10.26603/001c.73319. eCollection 2023. PMID 37020451
- [Background] Plisky P, Schwartkopf-Phifer K, Huebner B, Garner MB, Bullock G. Systematic Review and Meta-Analysis of the Y-Balance Test Lower Quarter: Reliability, Discriminant Validity, and Predictive Validity. Int J Sports Phys Ther. 2021 Oct 1;16(5):1190-1209. doi: 10.26603/001c.27634. eCollection 2021. PMID 34631241
- [Background] Powden CJ, Dodds TK, Gabriel EH. THE RELIABILITY OF THE STAR EXCURSION BALANCE TEST AND LOWER QUARTER Y-BALANCE TEST IN HEALTHY ADULTS: A SYSTEMATIC REVIEW. Int J Sports Phys Ther. 2019 Sep;14(5):683-694. PMID 31598406
- [Background] Smith E, Hoy DG, Cross M, Vos T, Naghavi M, Buchbinder R, Woolf AD, March L. The global burden of other musculoskeletal disorders: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis. 2014 Aug;73(8):1462-9. doi: 10.1136/annrheumdis-2013-204680. Epub 2014 Mar 3. PMID 24590181
- [Background] Taber JM, Leyva B, Persoskie A. Why do people avoid medical care? A qualitative study using national data. J Gen Intern Med. 2015 Mar;30(3):290-7. doi: 10.1007/s11606-014-3089-1. Epub 2014 Nov 12. PMID 25387439
- [Background] Teyhen DS, Rhon DI, Butler RJ, Shaffer SW, Goffar SL, McMillian DJ, Boyles RE, Kiesel KB, Plisky PJ. Association of Physical Inactivity, Weight, Smoking, and Prior Injury on Physical Performance in a Military Setting. J Athl Train. 2016 Nov;51(11):866-875. doi: 10.4085/1062-6050-51.6.02. Epub 2016 Oct 3. PMID 27690529
- [Background] Teyhen DS, Shaffer SW, Goffar SL, Kiesel K, Butler RJ, Rhon DI, Plisky PJ. Identification of Risk Factors Prospectively Associated With Musculoskeletal Injury in a Warrior Athlete Population. Sports Health. 2020 Nov/Dec;12(6):564-572. doi: 10.1177/1941738120902991. Epub 2020 Mar 5. PMID 32134698
- [Background] Yelin E, Weinstein S, King T. The burden of musculoskeletal diseases in the United States. Semin Arthritis Rheum. 2016 Dec;46(3):259-260. doi: 10.1016/j.semarthrit.2016.07.013. Epub 2016 Jul 26. No abstract available. PMID 27519477